CLINICAL TRIAL: NCT04723004
Title: A Randomized, Open-label, Multi-center Phase III Clinical Study to Evaluate the Safety and Efficacy of Toripalimab (JS001) Combined With Bevacizumab Versus Sorafenib as First-line Therapy for Advanced Hepatocellular Carcinoma
Brief Title: Evaluate the Safety and Efficacy of Toripalimab Combined With Bevacizumab Versus Sorafenib Therapy for HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JS001-035-III-HCC
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Toripalimab combined with Bevacizumab
  Interventions: Combination Product: Toripalimab combined with Bevacizumab
- Control group (Active Comparator): Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Combination Product: Toripalimab combined with Bevacizumab — Experimental group:
  Toripalimab, 240mg, IV infusion, every 3 weeks (q3w). combined with Bevacizumab 15mg/kg, IV infusion, every 3 weeks (q3w), Continuous infusion, in a cycle of 3 weeks (21 days), until occurrence of termination event specified in the protocol.
  Arms: Experimental group
Drug: Sorafenib — Control group:
  Sorafenib 400mg, po, Bid, continuous administration, until occurrence of termination event specified in the protocol.
  Arms: Control group

SUMMARY:
This is a prospective, randomized, open-label, parallel-group, active controlled, multi-center phase III registration clinical study to observe, compare and evaluate the efficacy and safety of Toripalimab (hereafter referred to as JS001) combined with Bevacizumab versus Sorafenib as the first-line therapy for advanced HCC This study will enroll the patients with locally advanced or metastatic hepatocellular carcinoma who could not be radically cured and not receive any prior systemic therapy. The study will use PFS and OS as the co-primary endpoints, with approximately 280 patients planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years (inclusive), male or female.
2. Histological or cytological diagnosis of HCC or clinical diagnosis of HCC in cirrhotic patients per the American Association for the Study of Liver Diseases (AASLD) guideline.
3. Unresectable BCLC B/C
4. No previous systemic therapy for HCC, patients with prior adjuvant therapy alone who relapsed at 6 months or above after the last adjuvant therapy may be enrolled.
5. ≥ 1 measurable lesion per RECISTv1.1.
6. Child-Pugh class A, with no history of hepatic encephalopathy.
7. ECOG PS 0 or 1.
8. Predicted life expectancy ≥12 weeks.
9. adequate main organ functions
10. In case of HBsAg (+) and/or HBcAb (+), HBV DNA is required to be < 2000 IU/mL. Patients with anti-HCV antibody positive and HCV- RNA>1000 copies/mL will be excluded; HBV/HCV co-infected patients will be excluded. patients with a prior history of HCV infection who tested negative for HCV-RNA can be considered HCV uninfected.
11. Female subjects of childbearing potential must receive serum pregnancy test within 7 days before randomization and the result should be negative, and should be willing to adopt reliable and effective contraceptive methods during the trial and within 60 days after the last dose of study drug. The male patients whose partners are women of childbearing potential must agree to use reliable and effective contraceptive methods during the trial and within 60 days after the last dose of study drug.
12. Being voluntary to participate in the study, sufficiently informed consent and signature of written informed consent form, with good compliance.

Exclusion Criteria：

1. Known ICC or mixed cell carcinoma, sarcomatoid HCC and hepatic fibrolamellar carcinoma.
2. History of malignancy other than HCC within 5 years prior to screening.
3. Hepatic surgery and/or local therapy or investigational treatment with for HCC within 4 weeks prior to randomization, or palliative radiotherapy for bone metastatic lesion within 2 weeks prior to randomization, or Chinese medicine preparation with anti-liver cancer effect within 2 weeks prior to randomization, and non-recovery (not recovered to ≤ NCI-CTCAE v5.0 grade 1) from side effects of any such treatment (except alopecia).
4. Prior other anti-PD-1 antibody therapy or other immunotherapy against PD- 1 / PD-L1.
5. Uncontrolled pericardial effusion, uncontrolled pleural effusion or clinically obvious moderate/severe pleural effusion at screening.
6. History of gastrointestinal hemorrhage within 6 months prior to randomization; the patients with portal hypertension need to receive gastroscopy to exclude the patients with "red sign", if they are considered by investigators to have high risk for hemorrhage (including moderate-to-severe esophageal and/or gastric varices with hemorrhagic risk, locally active peptic ulcer and persistent fecal occult blood (+)). The patient needs to be excluded if there is a history of "red sign" in gastroscopy.
7. Having ≥ grade 3 (NCI-CTC AE v5.0) gastrointestinal or non- gastrointestinal fistula at present.
8. Cancer thrombus in the main trunk of portal vein involving contralateral portal vein branch, or involving superior mesenteric vein. Cancer thrombus in inferior vena cava should be excluded.
9. Serious cardiovascular and cerebrovascular diseases
10. Having major bleeding and coagulation disorders or other obvious evidence on hemorrhagic tendency:
11. Medium to large surgical treatment within 4 weeks prior to randomization (except diagnostic biopsy).
12. Central nervous system metastases.
13. Serious, non-healing or dehiscing wound, active ulcer or untreated bone fracture.
14. Vaccination of live vaccine within 30 days prior to randomization.
15. Active autoimmune diseases requiring systemic treatment (i.e., immunomodulatory drug, corticosteroid or immunosuppressant) in the past 2 years; however, replacement therapy (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency), inhaled or topical corticosteroids will not be excluded.
16. History of clear interstitial lung disease or non-infectious pneumonia, unless induced by local radiotherapy; Presence of active tuberculosis during screening period or previous anti-tuberculosis treatment within one year prior to randomization.
17. Any serious acute and chronic infection requiring systemic antibacterial, antifungal or antiviral therapy at screening, not including viral hepatitis.
18. Known history of human immunodeficiency virus (HIV) infection.
19. Previously receiving allogeneic stem cell or solid organ transplantation.
20. Inability to swallow tablets, malabsorption syndrome or any condition that affects gastrointestinal absorption.
21. Known history of serious allergy to any monoclonal antibody, targeted anti- angiogenic drug.
22. Other unsuitable subjects as per the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  A duration from the date of initial treatment with Toripalimab Plus Bevacizumab or Sorafenib to disease progression (defined by RECIST 1.1) or death of any cause, whichever comes first.
Overall survival (OS) | Up to 2 years
  Duration from the date of initial treatment with Toripalimab Plus Bevacizumab or Sorafenib monotherapy to the date of death due to any cause.

SECONDARY OUTCOMES:
ORR | Up to 2 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
DoR | Up to 2 years
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Disease Control Rate (DCR) | Up to 2 years
  Proportion of patients with reduction and non-change in tumor burden of a predefined amount, including complete remission, partial remission and stable disease
TTP | Up to 2 years
  Define as the time from randomization to the first documented disease progression
Incidence of AEs/SAEs as Assessed by CTCAE v5.0 | From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years.
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
TMB | Up to 12 years
  Correlation between tumor mutation burden (TMB) and the efficacy of Toripalimab combined with Bevacizumab
ADA | Up to 12 years
  Serum levels and incidence of Anti-drug antibody of Toripalimab combined with Bevacizumab treatment group

CONTACTS AND LOCATIONS:
Locations (56):
- China (54):
  - The First Affiliated Hospital of Bengbu Medical college, Bengbu, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Southwest Hospital Of AMU, Chongqing, Chongqing Municipality
  - The Frist Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Wuwei Tumor Hospital, Wuwei, Gansu
  - The First Peoples Hospital of Foshan, Foshan, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - SSun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - he First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - NanJing Drum Tower Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The first Affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jilin Guowen Hospital, Changchun, Jilin
  - Liaoning cancer hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - Xi'an International Medical Center Hospital, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Gaoxiong, Taiwan
  - MacKay Memorial Hospital, Taibei, Taiwan
  - Changhua Christian Hospital, Zhanghua, Taiwan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - ShuLan（HangZhou) Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Tongji Hospital Tongji Medical College Of HUST, Wuhan, Zhejiang
  - Xiehe Hospital Tongji Medical College Of HUST, Wuhan, Zhejiang
  - Zhongnan Hospital of Wuhan University, Wuhan, Zhejiang
  - Jia Fan, Shanghai
- Singapore (2):
  - Curie Oncology, Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Derived] Shi Y, Han G, Zhou J, Shi X, Jia W, Cheng Y, Jin Y, Hua X, Wen T, Wu J, Gu S, Bai Y, Wang X, Zhang T, Chen Z, Zhang B, Huang M, Liu H, Mao Y, Zhou L, Wang R, Shan Y, Zhang W, Song T, Guo Y, Zhou F, Shao B, Zhang M, Liang B, Zheng J, Zhang G, Shen J, Su W, Zhang F, He Y, Hu S, Liu R, Zhang C, Shen S, Zeng H, Wang TE, Guo W, Shen Y, Chen Y, Li Y, Samol J, Hu H, Zhang W, Du C, Li E, Liu C, Pin CS, Li X, Xu H, Huang JF, Hao C, Lv J, Wang W, Xu Q, Bai A, Zhang X, Liu B, Jin C, Fan J. Toripalimab plus bevacizumab versus sorafenib as first-line treatment for advanced hepatocellular carcinoma (HEPATORCH): a randomised, open-label, phase 3 trial. Lancet Gastroenterol Hepatol. 2025 Jul;10(7):658-670. doi: 10.1016/S2468-1253(25)00059-7. Epub 2025 May 20. PMID 40409323